CLINICAL TRIAL: NCT05351372
Title: Low-dose Cone-beam Computed Tomography for Assessment of Alveolar Clefts, a Randomized Controlled Trial in Image Quality
Brief Title: Validation of X-ray Protocols in Cleft Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Tobias Regnstrand, Resident i Dentomaxillofacial radiology, PhD student, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 853386
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Evaluate CBCT Protocols in Subjective Image Quality
MeSH Terms: interventions — Clinical Protocols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ULD protocol (Experimental): ultra-low dose protocol in cone-beam computed tomography with a field of view including the cleft area
  Interventions: Radiation: Ultra-low dose protocol
- Standard dose protocol (Active Comparator): Standard dose protocol in cone-beam computed tomography with a field of view including the cleft area
  Interventions: Radiation: Standard dose protocol

INTERVENTIONS:
Radiation: Ultra-low dose protocol
  Arms: ULD protocol
Radiation: Standard dose protocol
  Arms: Standard dose protocol

SUMMARY:
Children born with an alveolar cleft receive bone grafts for improved function and aesthetics. The cleft area is radiologically examined before and post bone graft. Optimizing x-ray examination protocols is essential to protect these patients from possible delayed radiation injury later in life. This study investigates whether image quality of cone-beam computed tomography (CBCT) exposed with an ultra-low dose (ULD) protocol is comparable to the clinical default protocol, the standard dose (SD) protocol, in visualizing details of importance in bone grafting of alveolar clefts.

Methods In this randomized controlled study, 72 patients with uni- or bilateral alveolar clefts between 9-19 years (mean age 9.5) were randomized 1:1 with either a ULD or an SD CBCT examination protocol. The CBCT scans were conducted with Planmeca ProMax Mid with an 8x5cm field of view. Two experienced radiologists blindly evaluated the images and visibility of cortical bone border, trabecular bone, tooth anatomy, root development, periodontal space, and cleft width. The visibility was categorized as unacceptable, acceptable, or excellent.

DETAILED DESCRIPTION:
Radiographic imaging is an integral part of diagnostics, therapy planning and post-surgery assessment. Cone beam computed tomography (CBCT) was introduced in the late 90s and is now widely accepted. The technique utilizes a cone shaped X-ray beam to directly create a volumetric data, with predefined fields of view (FOV). CBCT provides 3D information with excellent spatial resolution, enabling assessment of anatomical variations and pathological changes in bone.

Cleft lip and palate disorder are among the most common birth defects, with the reported incidence in the Stockholm region of 1.7/1000 live births. The malformation can involve the lip, the alveolar process and the palate. When the alveolar process is involved CBCT can be indicated to assess the local anatomy prior to and after bone augmentation.

Minimizing the radiation dosage is especially important for children since the estimated risk for cancer formation or hereditable effects is approximately 3 times higher than for an adult aged 30.

Therefore the developments of low dose protocols within CBCT techniques are progressing rapidly. By applying more sensitive detector and a sophisticated image processing algorithm, the manufacturer Planmeca claimed that with Ultra Low Dose (ULD) protocol the effective patient dose may be reduced by up to 76%. A consequence of dramatically reduced exposure is the decreased signal-noise ratio, in other words reduced image quality, which results in increased diagnostic uncertainty of detailed structures. Since the accepted diagnostic image quality is highly associated with diagnostic tasks, clinical studies on evaluation new diagnostic feature are important.

HYPOTHESIS/RESEARCH QUESTION Will Promax 3D Mid CBCT with ULD normal dose protocol provide adequate information in order to assess necessary clinical questions in the region of the maxillary alveolar cleft compared to normal dose protocol?

METHODS Study design Randomized controlled trial examining the effect of two different Promax 3D Mid CBCT protocols, i.e. ULD normal dose setting versus normal dose setting, on image quality examining children with cleft involving the alveolar process.

Data source All patients with cleft involving the alveolar process, having treatment at Stockholm Craniofacial Centre Karolinska university hospital, being referred to Division of orofacial diagnostics and surgery - Image and functional odontology, Karolinska Institutet. Reason for referral CBCT examination to evaluate anatomy of the anterior maxilla prior to or after bone augmentation of the cleft located to the alveolar process.

Exposure/Intervention The exposure in the planned study is radiographic examination of children with cleft involving the alveolar process with CBCT Ultra Low Dose protocol compared with Normal dose protocol.

The study will be double blinded, nor will the patient nor the observers performing the evaluation of the images know the allocation. All observer assessment will be performed at one specific computer work station using the software program (Romexis Planmeca OY Helsinki Finland). The examinations will be executed by one of two possible nurses with extensive experience from handling CBCT devices. For the nurse the allocation cannot be concealed since the actual setting of the parameters has to be done manually. Therefore, a triple blinded design seems impossible. Since the same modality is used, Promax 3D Mid CBCT (Planmeca OY Helsinki Finland) for both protocols no evident risk exist that the patient or accompanying parent/guardian will work out the actual protocol in use.

In order to randomize the cases will be sectioned in groups of ten in a 1:1 assignment to either of the two protocols. The sequence for each group will be predetermined by lottery. Ten folded papers with equal size will be drawn by a person blindfolded without any knowledge of the study. The papers will be marked ULD for ULD normal dose protocol respectively NORMAL for normal dose protocol. The sequence for each group will be registered and provided up on the time for examination in a cover in the lab adjacent to the CBCT device. The idea with dividing cases and controls in groups, five of each resulting in a total of ten, is to ensure that the relation between the numbers of the two protocols is balanced.

The image conditions chosen for the Field of View (FOV) is 80mm in diameter and 50mm in height. The reason for not choosing a smaller, FOV i.e. 40 x 50 mm, decreasing the effective dose even further, is to provide information also on the contralateral side of the maxilla, a request from the surgeons giving important information needed during treatment planning. Normal clinical procedure using axial, coronal and sagital reconstructions of 1 mm thick slices will be used for the evaluation. Axial slices are according to standard in 3D imaging reconstructed parallel to the hard palate while paracoronal and parasagittal are perpendicular to the alveolar crest on the cleft side. All reconstructive work and imaging will be made in the software program Romexis (Planmeca OY Helsinki Finland). The examinations and reconstructions will be similar of those in a recent study from Finland in 2014.

Two dentomaxillofacial radiologists with profound knowledge and experience in assessing CBCT images will evaluate all radiographic 3D material. The 3D volumes will randomly be displayed using the same model of monitor (RadiForce MX191; EIZO, Hakusan, Japan), with a built-in digital imaging and communications in medicine setting. The radiographs will be evaluated under dimmed room light and a viewing distance of about 50 cm. The observers are allowed to adjust the window setting for light intensity and contrast according to their own preferences.

According to a three-point scale, the image quality will be assessed based on how well the observers can identify anatomical structures of interest prior to or post bone graft (unacceptable=1, acceptable=2, excellent=3). The landmarks of evaluation will be the cortical border of bone adjacent to the cleft, alveolar bone nearby the cleft, tooth anatomy of teeth adjacent to the cleft, root development, the periodontal space, and the width of the cleft. Possible motion artefacts presented in the CBCT images will be registered as minor or apparent. In case of a discrepancy between the two radiologists, the mean value of the observer's ratings is recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cleft involving the alveolar process undergoing treatment at Stockholm Craniofacial Centre
* Reason for referral is CBCT examination in order to evaluate anatomy of the anterior maxilla prior to or after bone augmentation of the cleft
* Patient/parent has given informed consent to participate in the study.

Exclusion Criteria:

* No informed consent is given. Those patients will be examined according to standard clinical procedures.
* Patients with a medical history of disorder/syndrome/chronic disease that will affect both the examination and the outcome.
* No CBCT examination of the cleft area.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Subjective image quality | 6 months
  unacceptable=1, acceptable=2, excellent=3

SECONDARY OUTCOMES:
cortical border of bone adjacent to the cleft | 6 months
  unacceptable=1, acceptable=2, excellent=3
alveolar bone nearby the cleft | 6 months
  unacceptable=1, acceptable=2, excellent=3
tooth anatomy of teeth adjacent to the cleft | 6 months
  unacceptable=1, acceptable=2, excellent=3
root development | 6 months
  unacceptable=1, acceptable=2, excellent=3
periorontal space visibility | 6 months
  unacceptable=1, acceptable=2, excellent=3
Width of the cleft | 6 months
  unacceptable=1, acceptable=2, excellent=3

CONTACTS AND LOCATIONS:
Overall Officials: Xie-qi Shi, PhD, Principal Investigator — University of Bergen
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No